CLINICAL TRIAL: NCT05498506
Title: Risk Factors for the Usage of ≥3 Linear Stapler Cartridges During Double Stapling Anastomosis in Laparoscopic Low Anterior Resection of Rectal Cancer
Brief Title: Multiple Firings in Double-stapled Colorectal Anastomosis
Status: Completed | Type: Observational
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Principal Investigator, Cai Zhenghao, Director, department of medical-engineering collaboration, Shanghai Minimally Invasive Surgery Center
Other Study IDs: MISC-DST
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple linear stapler firings during double stapling technique (DST) is associated with anastomotic leakage (AL) after laparoscopic low anterior resection (LAR). We aim to investigate the risk factors and then to develop a deep learning model to predict the usage of ≥3 linear stapler cartridges during DST anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* 1) carcinoma of rectum confirmed by histopathological evaluation;
* 2) tumor located in the mid-low rectum (less than 10cm from the anal verge);
* 3) performance of DST anastomosis;
* 4) pelvic MRI obtained within 14 days before surgery.

Exclusion Criteria:

* 1) other anastomotic techniques (e.g., trans-anal rectal excision);
* 2) Hartmann's operation or other procedures without anastomosis;
* 3) the number of linear stapler cartridges was not traceable in the operative report.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent Laparoscopic anterior resection for mid-low rectal cancer at Ruijin Hospital, Shanghai, People's Republic of China, between 2016 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
the number of linear stapler cartridges | during surgery
  the number of linear stapler cartridges used during DST anastomosis

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China